CLINICAL TRIAL: NCT05260450
Title: Laser Treatment of Toenail Onychomycosis With a 1064 nm Nd:YAG-laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Christian Bisp Sørensen, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210020
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Onychomycosis of Toenail

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Long-pulsed group) (Experimental): Nail clippings allocated to group A received laser treatment with a 1064 nm Nd:YAG-laser. They received one treatment with laser settings: pulse duration 10 ms, spot size 3 mm, fluence 40-50 J/cm2, number of laser pulses 100 /cm2.
  Interventions: Device: 1064 nm Nd:YAG-laser therapy
- Group B (Short-pulsed group) (Active Comparator): Nail clippings allocated to group B received laser treatment with a 1064 nm Nd:YAG-laser. They received one treatment with laser settings: pulse duration 0.3 ms, spot size 3 mm, fluence 40 J/cm2, number of laser pulses 100 /cm2.
  Interventions: Device: 1064 nm Nd:YAG-laser therapy

INTERVENTIONS:
Device: 1064 nm Nd:YAG-laser therapy — All interventions and mycological tests for each subject were performed over the course of one day.
  After subjects were included, toenails with a clinical suspicion of OM were tested for fungal infection by culture and microscopy. At the same time, nail clippings from said toenails were obtained and randomised into one of two treatment groups, i.e., group A and group B.
  The nail clippings were then treated with a 1064 nm Nd:YAG-laser with laser settings as specified by the treatment groups. All nail clippings were treated only once.
  Immediately after treatment, nail clippings were again tested for fungal infection by culture and microscopy.

SUMMARY:
This study aims to assess if laser treatment can cure fungal infection in toenails.

Nail clippings from eligible subjects were obtained and randomised into two groups. All nail clippings were treated once with a 1064 nm Nd:YAG-laser. Before and after treatment, nail clippings were tested for fungal infection by microscopy and by culture.

DETAILED DESCRIPTION:
This study was carried out as a randomised controlled trial (RCT) including two treatment groups subjected to two different laser treatments. A 1064 nm Nd:YAG-laser (Candela Medical, Ellipse Nordlys (Nd:YAG 1064), USA) was used for all treatments.

Potential subjects were recruited from general practitioners and skin clinics in North Jutland from August 24th, 2021, through December 2021.

All interventions and mycological tests for each subject were performed over the course of one day.

After subjects were included, toenails with a clinical suspicion of onychomycosis (OM) were tested for fungal infection by culture and microscopy. At the same time, nail clippings from said toenails were obtained and randomised into one of two treatment groups, i.e., group A and group B.

The nail clippings were then treated with a 1064 nm Nd:YAG-laser with laser settings as specified by the treatment groups. All nail clippings were treated only once.

Immediately after treatment, nail clippings were again tested for fungal infection by culture and microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years)
* Clinical suspicion of fungal infection in at least one toenail
* Signed informed consent
* Sufficient nail material to perform two cultures and one nail clipping

Exclusion Criteria:

* Administration of oral antifungal medication in the last 12 months or topical antifungal medication in the last month
* Diabetes mellitus with associated peripheral artery disease (PAD) or neuropathy
* Under the influence of alcohol or illegal narcotics
* Unable to understand written and spoken Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Fungal infection status in nail clippings measured by microscopy after laser treatment. | Approximately 10 minutes after treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by microscopy after therapy.
Fungal infection status in nail clippings measured by culture after laser treatment. | Approximately 10 minutes after treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by culture after therapy.
Fungal infection status in nail clippings measured by microscopy before laser treatment. | Approximately 10 minutes before treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by microscopy before therapy.
Fungal infection status in nail clippings measured by culture before laser treatment. | Approximately 10 minutes before treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by culture before therapy.

SECONDARY OUTCOMES:
Fungal infection status in nail clippings measured by PCR before laser treatment. | Approximately 10 minutes before treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by PCR before therapy.
Fungal infection status in nail clippings measured by PCR after laser treatment. | Approximately 10 minutes after treatment
  The number (rate) of included nail clippings in each group that were found negative for fungal infection measured by PCR after therapy.
Nail clippings temperatures | Approximately 2 seconds after end of treatment.
  Nail clippings temperature measured at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No